CLINICAL TRIAL: NCT01147796
Title: Accuracy of the 64 Slices Computed Tomography for the Diagnosis of Left Atrial Appendage Thrombus
Acronym: THROMBI-SCAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: defect of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P080607
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2013-09

CONDITIONS: Thrombus
Keywords: Thrombus; computed tomography; Transoesophageal echocardiography
MeSH Terms: conditions — Thrombosis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrombus (Active Comparator): patients with positive TEE (thrombus)
  Interventions: Device: computed tomography
- No thrombus (Placebo Comparator): patients with negative TEE (no thrombus)
  Interventions: Device: computed tomography

INTERVENTIONS:
Device: computed tomography — 64 slices CT with iodine injection
  Arms: Thrombus
Device: computed tomography — 64 slices CT with iodine injection
  Arms: No thrombus

SUMMARY:
Transoesophageal echocardiography (TEE) is considered as the gold standard method for detection of left atrial appendage (LAA) thrombus but is a semi-invasive investigation. The primary aim of the study is to evaluate the accuracy of the 64 slices CT using prospective gating for the diagnosis LAA thrombus. The secondary objective is to defined the optimal acquisition time offering the best diagnostic performance (early, late or both).

DETAILED DESCRIPTION:
Left atrial appendage (LAA) thrombus is a major cause of cardiogenic embolism. It is responsible of high morbidity and mortality and translates into significant modifications of patient management. Transoesophageal echocardiography (TEE) is considered as the gold standard method for detection of LAA thrombus but is a semi-invasive investigation. TEE is indeed performed using intravenous benzodiazepines sedation in order to optimize patient tolerance and quality for the operator or even under general anesthesia. To date there is no other validated method for the assessment of LAA thrombus. Multidetector computed tomography (CT) is currently widely used the assessment of cardiac function and geometry as well as coronary artery anatomy. Technologic improvement with the 64 slices CT, offering a high temporal and spatial resolution, and the new prospective gating, reducing drastically the irradiation dose, make it particularly attractive for the assessment of LAA thrombus but it has never been evaluated is this indication. Furthermore, the addition to the current arterial or "early" acquisition time, a second "late" acquisition (2 minutes later) may reduce false positive results.

Aims of the study. The primary aim of the study is to evaluate the accuracy of the 64 slices CT using prospective gating for the diagnosis LAA thrombus. The secondary objective is to defined the optimal acquisition time offering the best diagnostic performance (early, late or both).

Design of the study. The present study is a preliminary MONOCENTER study in which TEE is the reference method and the 64 slices CT with iodine injection and prospective gating the method to assess. All patients hospitalized at BICHAT hospital and referred for a TEE clinically motivated by search of a LAA thrombus are potential candidates for the present study. To insure the feasibility of the study with a rigorous methodology TEE will be performed in all patients but the prevalence of LAA thrombus will be deliberately increased and patients with negative TEE (no thrombus) to whom the CT will be performed will be randomized. Both TEE and CT will be performed within 18 hours. All CT analysis will be centralized and performed blinded of any clinical of echocardiographic information at the end of the inclusion period of the study. We planned to enroll 135 patients under a two years period.

Clinical implications. Validation of the 64 slices computed tomography with prospective gating may reduce TEE indications and improve patients' comfort.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized at BICHAT hospital and referred for a TEE clinically motivated by search of a LAA thrombus
* 18 years old
* signed informed consent 3 hours after TEE,
* Have health insurance.

Exclusion Criteria:

* woman into old of procreates
* impaired renal function
* Renal Hypoperfusion
* drugs nephrotoxic
* myeloma
* iodine injection 48 h before the inclusion
* over-sensitiveness with a product of iodized contrast
* Contra-indication for CT with iodine injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
diagnosis LAA thrombus | 24 h
  evaluate the accuracy of the 64 slices CT using prospective gating for the diagnosis LAA thrombus

SECONDARY OUTCOMES:
optimal acquisition time | 24H
  the optimal acquisition time offering the best diagnostic performance

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel : Serfaty, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat, Paris, France